CLINICAL TRIAL: NCT02863796
Title: The Safety and Feasibility of the WhiteSwell System for the Reduction of Interstitial Fluid Overload in Patients With Acutely Decompensated Heart Failure
Brief Title: Safety and Feasibility of the WhiteSwell System"
Acronym: SWIFTHF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: WhiteSwell, Limited (Industry)
Collaborators: Avania (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2016-001
Record Dates: First submitted 2016-07-06; First posted 2016-08-11 (Estimated); Last update posted 2022-04-19 (Actual); Status verified 2022-04

CONDITIONS: Heart Failure; Congestive Heart Failure
Keywords: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Single arm (Experimental): This prospective, multi-center, single arm study is designed to evaluate the safety and feasibility of the WhiteSwell System in the reduction of interstitial fluid overload in patients with acutely decompensated heart failure (ADHF)
  Interventions: Device: WhiteSwell System

INTERVENTIONS:
Device: WhiteSwell System — To promote movement of interstitial fluid to the intravascular space to allow for the body to remove it, in conjunction with a diuresis regimen.

SUMMARY:
Early feasibility study to evaluate safety and performance of the WhiteSwell System in the treatment of fluid overload in hospitalized patients with acutely decompensated heart failure.

DETAILED DESCRIPTION:
This study will evaluate the safety and feasibility of the WhiteSwell System for the treatment of patients hospitalized with acutely decompensated heart failure. Subjects who have been admitted to the hospital less than 72 hours for ADHF will be evaluated for inclusion into the study.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18
2. Subject is admitted to the hospital with a primary diagnosis of acute decompensated heart failure (ADHF).
3. Subjects receiving IV diuretic for ADHF and demonstrating fluid overload. This includes a minimum of 2 of the following:

   * peripheral edema ≥ +2 (on a 0 to +3 scale, indicating indentation of skin with mild digital pressure that requires 10 s or more to resolve in any dependent area including extremities or sacral region);
   * jugular venous distension ≥8 cm H2O
   * pulmonary edema or pleural effusion on chest radiograph
   * enlarged liver or ascites;
   * paroxysmal nocturnal dyspnea or ≥ two-pillow orthopnea;
   * dyspnea at rest with respiration rate ≥20 per minute
4. Renal function parameters: 30<eGFR<80
5. Biomarkers: BNP/pro-BNP

   1. BNP>400 pg/ml or NT-pro-BNP>1,600 pg/ml
   2. For patients with rate-controlled persistent or permanent AF: BNP>600 pg/ml or NT-pro-BNP>2,400 pg/ml
6. Subject must be able to be enrolled into the trial ≤ 72 hours of their admission to the hospital
7. Subject agrees to comply with all follow-up evaluations
8. Subject has provided written informed consent; or if unable to perform informed consent, written informed consent on behalf of the subject has been provided by a legally-authorized representative

Exclusion Criteria:

1. Subjects requiring inotropic therapy, mechanical ventilation, or mechanical circulatory support
2. Subjects developing worsening renal function (creatinine >0.5 mg/dL above baseline) within the time frame from admission to enrollment.
3. Subject has experienced a thromboembolic event (eg, pulmonary embolism (PE), deep vein thrombosis (DVT)) within the previous 6 months
4. Subject has contraindications to systemic anticoagulation
5. Subject with INR >1.8 or on novel anticoagulants (NOACs). Subjects who have taken NOACs may be enrolled if a minimum of 48 hours has passed since their last dose, with the exception of subjects on Dabigatran, who may not be enrolled.
6. Subject has mechanical heart valve.
7. Subject with systolic blood pressure < 90mmHg at time of enrollment
8. Subject has evidence of active infection
9. Subject has anatomical abnormalities and variations, or visualization of the insertion and deployment site does not enable safe venous access and device deployment as assessed by ultrasound
10. Subject vein diameters proximal and distal to the internal jugular/subclavian vein bifurcation in area of device placement less than 13.5mm and/or greater than 205mm.
11. Subject has experienced transient ischemic attack (TIA) events or cerebrovascular events (CVA) at previous 6 months
12. Subject with Acute coronary syndrome (ACS).
13. Subject with severe concomitant disease expected to prolong hospitalization or expected to cause death in ≤ 90 days
14. Subject is pregnant. Pregnancy confirmed by positive urine or serum test, or lactating mothers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2019-04-24 (Actual); Study Completion 2022-03-14 (Actual)

PRIMARY OUTCOMES:
The Rate of adjudicated device- or procedure-related Serious Adverse Events vents | 30 days
  The rate of adjudicated device- or procedure-related Serious Adverse Events (SAEs). All primary safety endpoints will be reported as-adjudicated by the designated Clinical Events Committee (CEC) during treatment and through the 30-day follow-up period.

OTHER OUTCOMES:
Evaluation of Worsening Heart Failure During Device Therapy | During WhiteSwell Treatment Procedure (up to 72 hours)
  Worsening heart failure during device therapy, defined as worsening signs and/or symptoms of HF requiring intensification of HF therapy, including need for intensification of intravenous therapy with inotropes or mechanical therapy (e.g., mechanical ventilation, circulatory support)
Global clinical outcome encompassing mortality, symptoms, and renal function | Through study completion, an average of 1 month
  Death through day 30;
Global clinical outcome encompassing mortality, symptoms, and renal function | Through study completion, an average of 1 month
  Rehospitalization for heart failure to Day 30
Global clinical outcome encompassing mortality, symptoms, and renal function | Through study completion, an average of 1 month
  Worsening renal function during device therapy (>0.5 mg/dL increase in creatinine above baseline)
Global clinical outcome encompassing mortality, symptoms, and renal function | Through study completion, an average of 1 month
  Improvement in dyspnea based on the 7-point Likert scale
Global clinical outcome encompassing mortality, symptoms, and renal function | Through study completion, an average of 1 month
  Change in BNP levels from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: William T. Abraham, MD, Principal Investigator — Ohio State University
Locations (2):
- United States (2):
  - Advocate Health/Edwards Heart Hospital, Naperville, Illinois
  - Ohio State University, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No